CLINICAL TRIAL: NCT00757237
Title: An Open-Label, Randomized, Phase 3 Trial to Evaluate the Efficacy and Safety of Aztreonam for Inhalation Solution (AZLI) Versus Tobramycin Inhalation Solution (TIS) in an Intermittent Aerosolized Antibiotic Regimen in Subjects With Cystic Fibrosis Followed by an Open-Label, Single Arm Extension (European Union [EU] Only)
Brief Title: Aztreonam for Inhalation Solution vs Tobramycin Inhalation Solution in Patients With Cystic Fibrosis & Pseudomonas Aeruginosa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Chiltern International Inc. (Industry); ClinPhone, Inc. (Industry); Covance (Industry)
Responsible Party: Mark Bresnik, MD/Medical Monitor, GSI
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-205-0110
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Results first posted 2011-07-04 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Cystic Fibrosis
Keywords: aztreonam lysine; tobramycin inhalation solution; tobramycin nebuliser solution; cystic fibrosis; pseudomonas aeruginosa; lung infection; CFQ-R; inhaled antibiotic
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Aztreonam; Tobramycin; 2-(4-toluidino)-6-naphthalenesulfonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZLI 75 mg 3 times a day (TID) (Experimental)
  Interventions: Drug: Aztreonam for Inhalation Solution (AZLI)
- TIS 300 mg 2 times a day (BID) (Active Comparator)
  Interventions: Drug: Tobramycin Inhalation Solution (TIS)

INTERVENTIONS:
Drug: Aztreonam for Inhalation Solution (AZLI) — Aztreonam for inhalation solution (75 mg) was administered 3 times a day (TID) for 28 days for each treatment cycle via the PARI eFlow electronic nebulizer.
  Other Names: aztreonam; AZLI; inhaled antibiotic
  Arms: AZLI 75 mg 3 times a day (TID)
Drug: Tobramycin Inhalation Solution (TIS) — Tobramycin inhalation solution (300 mg) was administered 2 times a day (BID) for 28 days for each treatment cycle via the PARI LC Plus nebulizer with compressor or via another nebulizer compatible with country-specified labeling.
  Other Names: tobramycin; TNS; inhaled antibiotic
  Arms: TIS 300 mg 2 times a day (BID)

SUMMARY:
The purpose of this study was to assess the comparative safety and effectiveness of aztreonam for inhalation solution versus tobramycin inhalation solution in adult and pediatric patients with cystic fibrosis (CF) and pulmonary Pseudomonas aeruginosa (PA) infection.

DETAILED DESCRIPTION:
Number of Subjects Planned: Approximately 240 randomized patients

Target Population: CF patients >= 6 years of age with stable pulmonary disease, who at study entry had a recent positive sputum culture for PA and had been previously treated with aerosolized antibiotics without demonstration of drug intolerance.

The randomized phase of this study, used for hypotheses testing, enrolled participants from both the United States (US) and EU. An open-label, single-arm extension was available for participants in the EU who completed at least one course of AZLI or TIS during the randomized portion of the study. These participants were eligible to receive 3 additional cycles of AZLI in a 28-day, intermittent, repeating treatment regimen. Results of the extension phase will be available the first quarter (Q1) of 2012.

Randomized Phase Study Design (US and EU): This was an open-label, multicenter, randomized, parallel group study. The study design consisted of 2 treatment arms of 28-day, intermittent, repeating treatment regimens: aztreonam for inhalation solution (AZLI) or tobramycin inhalation solution (TIS). The total study period was 26 weeks. The study schedule included 9 visits - Screening, Baseline, Day 14, Day 28, followed by visits every 28 days through the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 6 years and older
* Subjects with CF as diagnosed by one of the following: documented sweat chloride >= 60 mEq/L by quantitative pilocarpine iontophoresis test, or documented sweat sodium >= 60 mmol/L, or 2 well characterized genetic mutations in the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) gene, or abnormal nasal potential difference with accompanying symptoms characteristic of CF
* Documented PA in an expectorated sputum or throat swab culture within 3 months prior to Visit 1 or at Visit 1
* Subjects must be able to provide written informed consent/assent prior to any study related procedures; parent/guardian must be able to give written informed consent as necessary prior to any study related procedure
* Subjects must have received previous treatment with aerosolized antibiotics without demonstration of drug intolerance
* FEV1 <= 75% predicted at Visit 1
* Ability to perform reproducible pulmonary function tests
* Chest radiograph at Visit 1 without significant acute findings (eg, infiltrates [lobar or diffuse interstitial], pleural effusion, pneumothorax); or chest radiograph or magnetic resonance image (MRI) obtained within the 180 days prior to Visit 1 without acute findings and no significant intercurrent illness; chronic, stable findings (eg, chronic scarring or atelectasis) are allowed

Exclusion Criteria:

* Current use of oral corticosteroids in doses exceeding the equivalent of 10 mg prednisone a day or 20 mg prednisone every other day
* History of sputum or throat swab culture yielding B. cepacia in the previous 2 years
* Current requirement for daily continuous oxygen supplementation or requirement for more than 2 L/minute at night
* Administration of any investigational drug or device within 28 days of Visit 1 or within 6 half-lives of the investigational drug (whichever is longer)
* Known local or systemic hypersensitivity to monobactam antibiotics
* Known allergies/intolerance to tobramycin
* Inability to tolerate inhalation of a short acting beta agonist
* Changes in or initiation of chronic azithromycin treatment within 28 days prior to Visit 1
* Administration of antipseudomonal antibiotics by inhalation, intravenous or oral routes within the 14 days prior to Randomization/Visit 2
* Changes in antimicrobial, bronchodilator (BD), dornase alfa, or corticosteroid medications within 7 days prior to Visit 1
* Changes in physiotherapy technique or schedule within 7 days prior to Visit 1
* History of lung transplantation
* Abnormal renal or hepatic function or serum chemistry at Visit 1, defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 5 times upper limit of normal range (ULN) or creatinine > 2 times ULN
* Positive pregnancy test at Visit 1; all women of childbearing potential will be tested
* Female of childbearing potential who is lactating or is not (in the opinion of the investigator) practicing an acceptable method of birth control; female subjects who utilize hormonal contraceptives as one of their birth control methods must have used the same method for at least 3 months before study dosing
* Any serious or active medical or psychiatric illness, which in the opinion of the investigator, would interfere with patient treatment, assessment, or compliance with the protocol

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bresnik, MD, Study Director — Gilead Sciences
Locations (80):
- United States (28):
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Tuscon, Arizona
  - Orange, California
  - Aurora, Colorado
  - Denver, Colorado
  - Wilmington, Delaware
  - Orlando, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Glenview, Illinois
  - Niles, Illinois
  - Boston, Massachusetts
  - Columbia, Missouri
  - Las Vegas, Nevada
  - Albany, New York
  - New Hyde Park, New York
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
- Austria (2):
  - Innsbruck
  - Salzburg
- Belgium (4):
  - Antwerp
  - Brussels
  - Ghent
  - Leuven
- Copenhagen, Denmark
- France (11):
  - Amiens
  - Bordeaux
  - Caen
  - Créteil
  - Lille
  - Lisieux
  - Montpellier
  - Nice
  - Paris
  - Pessac
  - Rennes
- Germany (9):
  - Berlin
  - Bochum
  - Essen
  - Giessen
  - Hamburg
  - Leipzig
  - Magdeburg
  - Mainz
  - München
- Ireland (2):
  - Dublin
  - Galway
- Italy (8):
  - Ancona
  - Catania
  - Milan
  - Napoli
  - Palermo
  - Parma
  - Rome
  - Verona
- Netherlands (2):
  - Maastricht
  - The Hague
- Portugal (2):
  - Lisbon
  - Porto
- Spain (2):
  - Madrid
  - Málaga
- Zurich, Switzerland
- United Kingdom (8):
  - Sheffield, West Yorkshire
  - Belfast
  - Cambridge
  - Cardiff
  - Leeds
  - Liverpool
  - London
  - Southampton

REFERENCES:
- [Derived] Assael BM, Pressler T, Bilton D, Fayon M, Fischer R, Chiron R, LaRosa M, Knoop C, McElvaney N, Lewis SA, Bresnik M, Montgomery AB, Oermann CM; AZLI Active Comparator Study Group. Inhaled aztreonam lysine vs. inhaled tobramycin in cystic fibrosis: a comparative efficacy trial. J Cyst Fibros. 2013 Mar;12(2):130-40. doi: 10.1016/j.jcf.2012.07.006. Epub 2012 Sep 15. PMID 22985692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy-three sites in the United States (US) and European Union (EU) enrolled a total of 274 participants in the study.
Pre-assignment Details: Of the 274 participants enrolled in the study, 273 were randomized between 07 August 2008 and 12 November 2009. One subject experienced a serious adverse event (SAE) between Visits 1 and 2; this subject did not receive study drug. A total of 268 participants received study drug (136 AZLI; 132 TIS).
Groups:
- AZLI (75 mg TID): AZLI (75 mg/1 mL aztreonam lysine when reconstituted in diluent [0.17% saline]; sterile, pH 4.2 to 7.0, and osmolality 300 to 550 mOsmol/kg). AZLI was self-administered by inhalation three times a day (TID) for 28 days for each treatment cycle using the investigational nebulizer.
- TIS (300 mg BID): TIS (300 mg/5 mL) was self-administered by inhalation two times a day (BID) for 28 days for each treatment cycle using the PARI LC PLUS(TM) Nebulizer with Compressor.
Period: Overall Study
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Started | 137 | 136
Treated | 136 | 132
Completed | 124 | 111
Not Completed | 13 | 25
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 8 | 12
Not completed — Safety or Tolerability | 3 | 5
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID) | Total
Number analyzed (Participants) | 136 | 132 | 268
Age Categorical [Number; unit: participants]
  >= 6 years to <= 12 years | 8 | 5 | 13
  > 12 years to < 18 years | 20 | 26 | 46
  >= 18 years | 108 | 101 | 209
Age Continuous [Mean (Standard Deviation); unit: years] | 25.8 (9.1) | 25.1 (9.0) | 25.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 66 | 134
  Male | 68 | 66 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 130 | 131 | 261
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 44 | 50 | 94
  Europe | 92 | 82 | 174
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 20.22 (2.95) | 20.49 (2.82) | 20.35 (2.88)
Inhaled Tobramycin Use in the Previous 12 Months [Number; unit: participants]
  < 84 days | 21 | 19 | 40
  >= 84 days | 115 | 113 | 228
Disease Severity [Number; unit: participants] — Forced Expiratory Volume (FEV1) percent predicted is a normalized value of FEV1 calculated using the Knudson equation and based upon participant age, gender, and height. This baseline measure indicates the number of participants with FEV1 greater than 50% and less than or equal to 50% of the predicted value based on age, gender, and height at screening.
  participants
    <= 50% predicted | 60 | 57 | 117
    > 50% predicted | 76 | 75 | 151
Forced Expiratory Volume (FEV1) Percent Predicted [Mean (Standard Deviation); unit: percent] — FEV1 percent predicted is a normalized value of FEV1 calculated using the Knudson equation and based upon participant age, gender, and height.
  percent | 52.30 (15.56) | 52.24 (14.57) | 52.27 (15.06)
Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Symptoms Scale (RSS) Score [Mean (Standard Deviation); unit: units on a scale] — The CFQ-R is a validated, patient-reported outcome tool measuring health-related quality of life for children and adults with CF. The CFQ-R contains both general and CF-specific scales. Respiratory symptoms (e.g., coughing, congestion, wheezing) are assessed with the CFQ-R Respiratory Symptoms Scale (RSS). The range of scores (units) is 0 to 100 with higher scores indicating fewer symptoms.
  units on a scale | 62.87 (20.42) | 58.02 (20.76) | 60.44 (20.69)

OUTCOME MEASURES:

1. Primary Outcome: Relative Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Percent Predicted at Day 28
Description: Spirometry was performed according to American Thoracic Society (ATS) guidelines at each visit. FEV1 percent predicted is a normalized value of FEV1 calculated using the Knudson equation and based upon participant age, gender, and height. Treatment effect on the relative change from baseline in FEV1 percent predicted at Day 28 (Visit 4) was tested using an analysis of covariance (ANCOVA) model-based method.
Time Frame: Baseline and end of treatment Course 1 (Day 28)
Population: Analysis was based on ITT population (all participants randomized to treatment who received at least part of one dose of study drug). The last observation carried forward (LOCF) method was used to impute missing data.
Measure: Least Squares Mean (Standard Error); unit: percent change in FEV1 percent predicted
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 136 | 132
percent change in FEV1 percent predicted | 8.35 (1.70) | 0.55 (1.77)
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: AZLI was inferior to TIS by more than 4% in the mean relative change of FEV1 percent predicted at Day 28. With 120 subjects per treatment group there was at least 85% power to declare noninferiority based on relative change from baseline at Day 28 in FEV1 percent predicted using the upper bound of a 2-tailed 95% CI for the difference in means with a noninferiority margin of 4, assuming a common standard deviation of 18% and true difference in means [TIS-AZLI] of -3.2%; Test type: Non-Inferiority or Equivalence — The treatment difference (TIS-AZLI) and standard error from the ANCOVA model were used to compute the two-sided 95% confidence interval. If the 95% upper boundary was less than the pre-specified non-inferiority margin of 4%, then the null hypothesis was rejected; p = 0.0001, ANCOVA — Based on the Benjamini & Hochberg method, non-inferiority at Day 28 for relative change in FEV1 percent predicted was assessed at the 0.05 level, given the significance of the coprimary endpoint (p<0.05); ANCOVA model included treatment, Day 0 FEV1 percent predicted, and previous inhaled tobramycin use for all participants; Mean Difference (Final Values) = -7.80, 95% CI 2-sided [-11.73 to -3.86] — Treatment difference refers to TIS-AZLI

2. Primary Outcome: Mean Actual Change From Baseline in FEV1 Percent Predicted Across 3 Treatment Courses
Description: Spirometry was performed according to ATS guidelines at each visit. FEV1 percent predicted is a normalized value of FEV1 calculated using the Knudson equation and based upon participant age, gender, and height.
  Treatment effect on the average adjusted means for the actual change in FEV1 percent predicted at Visits 4, 6, and 8 (Weeks 4, 12, and 20) was tested by mixed-effect model repeated measures (MMRM) analysis using the ITT population analysis set.
Time Frame: Baseline, and end of treatment Courses 1 (Week 4), 2 (Week 12), and 3 (Week 20)
Population: Analysis was based on ITT population (all participants randomized to treatment who received at least part of one dose of study drug).
Measure: Least Squares Mean (Standard Error); unit: actual change in FEV1 percent predicted
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 136 | 132
actual change in FEV1 percent predicted | 2.05 (0.69) | -0.66 (0.72)
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: there was no difference between AZLI and TIS treatment groups in the mean actual change of FEV1 percent predicted across 3 treatment courses among all participants. With 120 subjects per treatment group, there was at least 90% power at a 5% significance level to detect differences based upon actual change from baseline in FEV1 percent predicted (3.61%, 2.98%, 2.32%) between AZLI and TIS at Weeks 4, 12, and 20 with a common standard deviation of 9%; Test type: Superiority or Other; p = 0.0023, MMRM analysis — Based on the Benjamini & Hochberg method, superiority at Weeks 4, 12, and 20 of actual change in FEV1 percent predicted was tested at the 0.05 level, given the significance of the coprimary endpoint (p<0.05); MMRM analysis included Day 0 FEV1 percent predicted, previous inhaled tobramycin use, treatment, visit, and treatment/visit interaction; Mean Difference (Final Values) = -2.70 — Treatment difference refers to TIS-AZLI

3. Secondary Outcome: Relative Change From Baseline in FEV1 Percent Predicted at Day 28 in Subjects Who Received Inhaled Tobramycin for >= 84 Days in the 12 Months Prior to Randomization
Description: Spirometry was performed according to ATS guidelines. FEV1 percent predicted is a normalized value of FEV1 calculated using the Knudson equation and based upon participant age, gender, and height. Treatment effect on the relative change from baseline in FEV1 percent predicted at Day 28 (Visit 4) was tested using an ANCOVA model-based method, using the population of participants with prior inhaled tobramycin use of >= 84 days in the previous 12 months.
Time Frame: Baseline and end of treatment Course 1 (Day 28)
Population: Analysis was based on participants with previous inhaled tobramycin use of >= 84 days within the previous 12 months using the ITT analysis set. The last observation carried forward (LOCF) method was used to impute missing data for statistical analyses.
Measure: Least Squares Mean (Standard Error); unit: percent change in FEV1 percent predicted
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 115 | 113
percent change in FEV1 percent predicted | 10.04 (1.56) | 0.54 (1.57)
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: AZLI was inferior to TIS by more than 4% in terms of the participant means in relative change of FEV1 percent predicted at Day 28 among all participants having >= 84 days of inhaled tobramycin use in the previous 12 months; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.0001, ANCOVA — Secondary endpoints were tested sequentially by the closed testing procedure initiated by the significance of the primary endpoints. Given the coprimary endpoints were met at the 0.05 level, this non-inferiority endpoint was tested at the 0.05 level; ANCOVA model included treatment and Day 0 FEV1 percent predicted; Mean Difference (Final Values) = -9.50, 95% CI 2-sided [-13.86 to -5.14] — Treatment difference refers to TIS-AZLI

4. Secondary Outcome: Mean Actual Change From Baseline in FEV1 Percent Predicted Across 3 Treatment Courses in Subjects Who Received Inhaled Tobramycin for >= 84 Days in the 12 Months Prior to Randomization
Description: Spirometry was performed according to ATS guidelines at each visit. FEV1 percent predicted is a normalized value of FEV1 calculated using the Knudson equation and based upon participant age, gender, and height.
  Treatment effect on the average adjusted means for the actual change in FEV1 percent predicted at Visits 4, 6, and 8 (Weeks 4, 12, and 20) was tested by MMRM analysis using the population of participants with prior inhaled tobramycin use of >=84 days in the previous 12 months.
Time Frame: Baseline and end of treatment Courses 1 (Week 4), 2 (Week 12), and 3 (Week 20)
Population: Analysis was based on participants with prior inhaled tobramycin use >= 84 days in the previous 12 months using the ITT analysis set.
Measure: Least Squares Mean (Standard Error); unit: actual change in FEV1 percent predicted
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 115 | 113
actual change in FEV1 percent predicted | 3.26 (0.65) | -0.21 (0.66)
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: there was no difference between AZLI and TIS treatment groups in the mean actual change of FEV1 percent predicted across 3 treatment courses in the stratum of subjects having >=84 days of inhaled tobramycin use in the previous 12 months; Test type: Superiority or Other; p = 0.0002, MMRM analysis — Secondary endpoints were tested sequentially to control the Type I error rate based on the closed testing procedure. Given the significance of the coprimary endpoints and previous secondary endpoint, this endpoint was also tested at the 0.05 level; MMRM analysis included treatment, Day 0 FEV1 percent predicted, visit, treatment, and treatment/visit interaction for all participants; Mean Difference (Final Values) = -3.47 — Treatment difference refers to TIS-AZLI

5. Secondary Outcome: Time to Need for Intravenous (IV) Antipseudomonal Antibiotics for Respiratory Events
Description: IV antipseudomonal antibiotic use for a respiratory event was determined through the adjudication of events by a sponsor-independent, blinded review committee.
  Use was compiled from data recorded on the concomitant medications electronic case report form (eCRF) and compared to reported adverse events (AEs) to determine use for a respiratory event. The time to IV antipseudomonal antibiotic use was measured in days from baseline (Visit 2) to the date of first IV antipseudomonal antibiotic use or the date of study completion (last visit)/or early withdrawal if censored.
Time Frame: Day 0 to Day 168 (end of study)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 136 | 132
days | NA [177 to NA] — NA = Not estimable; less than 50% of the participants had an event by the end of the study. | 151 [113 to NA] — NA = Not estimable; less than 50% of the participants had an event by the end of the study.
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: there was no difference between AZLI and TIS treatment groups with respect to time to need for IV antipseudomonal antibiotics for respiratory events; Test type: Superiority or Other; p = 0.0025, Log Rank — [p-value comment as in outcome 4, analysis 1]

6. Secondary Outcome: Time to First Respiratory Hospitalization
Description: This endpoint was determined through the adjudication of events by a sponsor-independent, blinded review committee. Committee members reviewed all hospitalizations and determined which were related to respiratory events.
  Details of all hospitalizations, including the dates of admission and discharge, were recorded on the serious adverse event (SAE) eCRF.
  Time to first respiratory hospitalization was the number of days from baseline (Visit 2) to the date of first respiratory hospitalization or the date of study completion (last visit) /or early withdrawal if censored.
Time Frame: Day 0 to Day 168 (end of study)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 136 | 132
days | NA [NA to NA] — NA = Not estimable; less than 50% of the participants had an event by the end of the study. | NA [NA to NA] — NA = Not estimable; less than 50% of the participants had an event by the end of the study.
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: there was no difference between AZLI and TIS treatment groups with respect to time to first respiratory hospitalization; Test type: Superiority or Other; p = 0.1114, Log Rank — [p-value comment as in outcome 4, analysis 1]

7. Other Pre Specified Outcome: Actual Change From Baseline in CF Questionnaire - Revised (CFQ-R) Respiratory Symptoms Scale (RSS) Score at Day 28
Description: The CFQ-R is a validated patient-reported outcome tool measuring health-related quality of life for children and adults with CF. The CFQ-R contains both general and CF-specific scales. The endpoint was change in respiratory symptoms (e.g., coughing, congestion, wheezing) from baseline, assessed with the CFQ-R RSS (range of scores [units]: 0-100; higher scores indicate fewer symptoms).
Time Frame: Baseline and end of treatment Course 1 (Day 28)
Population: Analysis was based on ITT population (all participants randomized to treatment who received at least part of one dose of study drug). LOCF method was used to impute missing data for statistical analyses.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 136 | 132
Units on a scale | 8.20 (1.68) | 2.59 (1.73)
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: there was no difference between AZLI and TIS treatment groups in change from baseline in CFQ-R RSS scores at Day 28; Test type: Superiority or Other; p = 0.0048, ANCOVA — No adjustments were made for multiple comparisons; ANCOVA model included treatment, Day 0 FEV1 percent predicted, Day 0 CFQ-R RSS score, and previous inhaled tobramycin use; Mean Difference (Final Values) = -5.61 — Treatment difference refers to TIS-AZLI

8. Other Pre Specified Outcome: Mean Actual Change From Baseline in CFQ-R RSS Score Across 3 Treatment Courses
Description: The CFQ-R is a validated patient-reported outcome tool measuring health-related quality of life for children and adults with CF. The CFQ-R contains both general and CF-specific scales. The endpoint was the average actual change in respiratory symptoms (e.g., coughing, congestion, wheezing) from baseline, assessed with the CFQ-R RSS (range of scores [units]: 0-100; higher scores indicate fewer symptoms) at the end of each treatment course (Weeks 4, 12, and 20).
Time Frame: Baseline and end of treatment Courses 1 (Week 4), 2 (Week 12), and 3 (Week 20)
Population: Analysis was based on ITT population (all participants randomized to treatment who received at least part of one dose of study drug). The LOCF method was used to impute missing data for statistical purposes.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 136 | 132
units on a scale | 6.30 (1.49) | 2.17 (1.54)
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: there was no difference between AZLI and TIS treatment groups in the average actual change in respiratory symptoms at the end of each treatment course (Weeks 4, 12, and 20); Test type: Superiority or Other; p = 0.0189, ANCOVA — No adjustments were made for multiple comparisons; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -4.13 — Treatment difference refers to TIS-AZLI

9. Other Pre Specified Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) - Global Satisfaction Results at Week 20
Description: This 14 item questionnaire consists of 3 subscales that gauge participant perceptions of a medication's effectiveness, side effects, and convenience. The measure also contains a global satisfaction scale to evaluate overall participant satisfaction. The global satisfaction score is the endpoint reported here. The range of scores is 0 to 100, with higher scores indicating greater satisfaction.
Time Frame: At Week 20
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 130 | 126
units on a scale | 75.85 (4.58) | 61.73 (4.90)
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: there was no difference between AZLI and TIS treatment groups in the global satisfaction results of the TSQM at Week 20 (Day 140); Test type: Superiority or Other; p = 0.0097, ANCOVA — No adjustments were made for multiple comparisons; ANCOVA model included treatment, Day 0 FEV1 percent predicted, and previous inhaled tobramycin use; Mean Difference (Final Values) = -14.12 — Treatment difference refers to TIS-AZLI

10. Other Pre Specified Outcome: Total Number of Respiratory Hospitalizations
Description: Respiratory hospitalizations were determined through the adjudication of events by a sponsor-independent, blinded review committee. Committee members reviewed hospitalizations and determined which were related to respiratory events.
Time Frame: Day 0 to Day 168 (end of study)
Population: as for outcome 2
Measure: Number; unit: hospitalizations
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 136 | 132
hospitalizations | 40 | 58
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: there was no difference between AZLI and TIS treatment groups in the total number of respiratory hospitalizations from Day 0 to Day 168 (end of study); Test type: Superiority or Other; p = 0.044, negative binomial regression method — No adjustments were made for multiple comparisons

11. Other Pre Specified Outcome: Number of Respiratory Events Requiring IV and/or Inhaled Antipseudomonal Antibiotics (Other Than Randomized Treatment)
Description: Inhaled and/or IV antipseudomonal antibiotic use for respiratory event was determined through event adjudication by a sponsor-independent, blinded review committee. Use of IV and/or inhaled antipseudomonal antibiotics was compiled from data recorded on the concomitant medications eCRF and compared to reported AEs to determine use for a respiratory event. The time to IV and/or inhaled antipseudomonal antibiotic use was measured in days from baseline (Visit 2) to the date of first antipseudomonal antibiotic use or the date of study completion (last visit)/or early withdrawal if censored.
Time Frame: Day 0 through Day 168 (end of study)
Population: as for outcome 2
Measure: Number; unit: events
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 136 | 132
events | 84 | 121
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: there was no difference between AZLI and TIS treatment groups in the total number of respiratory events requiring IV and/or inhaled antipseudomonal antibiotics (other than randomized treatment) from Day 0 to Day 168 (end of study); Test type: Superiority or Other; p = 0.004, negative binomial regression method — No adjustments were made for multiple comparisons

12. Other Pre Specified Outcome: Time to Need for Inhaled and/or IV Antipseudomonal Antibiotics for Respiratory Event (Other Than Randomized Treatment)
Description: Antipseudomonal antibiotic use for respiratory event was determined through event adjudication by a sponsor-independent, blinded review committee.
  Use of IV and/or inhaled antibiotics for a respiratory event was compiled from data recorded on the concomitant medications eCRF and compared to reported AEs to determine use for a respiratory event. The time to antibiotic use for a respiratory event was measured in days from baseline (Day 0) to the date of first antibiotic use for a respiratory event or the date of study completion (last visit)/or early withdrawal if censored.
Time Frame: Day 0 to Day 168 (end of study)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Number analyzed (Participants) | 136 | 132
days | NA [177 to NA] — NA = Not estimable; less than 50% of the participants had an event by the end of the study. | 117 [102 to 169]
Statistical Analysis 1: Comparison: AZLI (75 mg TID) vs TIS (300 mg BID); Null hypothesis: there was no difference between AZLI and TIS treatment groups with respect to time to need for inhaled and/or IV antipseudomonal antibiotics for respiratory events; Test type: Superiority or Other; p = 0.0004, Log Rank — No adjustments were made for multiple comparisons

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AEs) were collected continuously from Day 0 (first dose) through Day 168 (Week 24).
Description: An AE was any physical/clinical worsening in symptoms/disease (including clinically significant change in lab values) experienced by a participant at any time during study, whether or not the AE was considered related to study participation or procedures. Participants were only counted once within a System Organ Class (SOC) and preferred term.
Arm/Group | AZLI (75 mg TID) | TIS (300 mg BID)
Serious Adverse Events (participants affected / at risk) | 42/136 | 44/132
Other Adverse Events (participants affected / at risk) | 128/136 | 127/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZLI (75 mg TID) (N=136) | TIS (300 mg BID) (N=132)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Distention (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 1 (1)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Body Temperature Increased (Investigations) | 0 (0) | 1 (1)
Breath Sounds Abnormal (Investigations) | 1 (1) | 1 (1)
C-Reactive Protein Increased (Investigations) | 1 (1) | 0 (0)
Catheter Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 3 (3) | 2 (2)
Chills (General disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (31) | 26 (30)
Cyanosis (Cardiac disorders) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (13) | 15 (17)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Exercise Tolerance Decreased (General disorders) | 6 (6) | 3 (3)
Fatigue (General disorders) | 1 (1) | 3 (3)
Feeding Tube Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forced Expiratory Volume Decreased (Investigations) | 3 (3) | 0 (0)
Glycosylated Haemoglobin Increased (Investigations) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (4)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hyperaemia (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (2) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 1 (2)
Pain (General disorders) | 2 (2) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Poor Quality Sleep (Nervous system disorders) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 16 (21) | 23 (29)
Pulmonary Function Test Decreased (Investigations) | 5 (5) | 4 (4)
Pyrexia (General disorders) | 11 (13) | 8 (10)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Headache (Nervous system disorders) | 1 (1) | 0 (0)
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Systemic Candida (Infections and infestations) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Vein Disorder (Vascular disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZLI (75 mg TID) (N=136) | TIS (300 mg BID) (N=132)
Abdominal Pain (Gastrointestinal disorders) | 15 | 8
Arthalgia (Musculoskeletal and connective tissue disorders) | 10 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Breath Sounds Abnormal (Investigations) | 7 | 14
Chest Discomfort (General disorders) | 13 | 13
Chest Pain (General disorders) | 6 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 92 | 95
Decreased Appetite (Metabolism and nutrition disorders) | 17 | 17
Diarrhoea (Gastrointestinal disorders) | 4 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 28
Exercise Tolerance Decreased (General disorders) | 20 | 24
Fatigue (General disorders) | 23 | 22
Forced Expiratory Volume Decreased (Investigations) | 7 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 30 | 20
Headache (Nervous system disorders) | 28 | 27
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 6
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 29 | 26
Nausea (Gastrointestinal disorders) | 13 | 10
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 34 | 37
Pain (General disorders) | 9 | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 63 | 67
Pulmonary Function Test Decreased (Investigations) | 6 | 15
Pyrexia (General disorders) | 34 | 36
Rales (Respiratory, thoracic and mediastinal disorders) | 29 | 32
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 15 | 16
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 24 | 33
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Vomiting (Gastrointestinal disorders) | 12 | 14
Wheezing (Respiratory, thoracic and mediastinal disorders) | 13 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or

The study has been completed at all study sites for at least 2 years.